CLINICAL TRIAL: NCT04089150
Title: MASTERPLAN: A Randomised Phase II Study of MFOLFIRINOX And Stereotactic Radiotherapy (SBRT) for Pancreatic Cancer With High Risk and Locally Advanced Disease
Brief Title: MFOLFIRINOX And Stereotactic Radiotherapy (SBRT) for Pancreatic Cancer With High Risk and Locally Advanced Disease
Acronym: MASTERPLAN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: Trans Tasman Radiation Oncology Group (Other); Australian Government Department of Health and Ageing (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC 0245/AGITG AG0118PS
Record Dates: First submitted 2019-02-04; First posted 2019-09-13 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Pancreatic Cancer
Keywords: stereotactic body radiotherapy; SBRT; chemotherapy; radiotherapy; surgery
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Leucovorin; Irinotecan; Fluorouracil; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Capecitabine; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): * Option 1: fluorouracil(5-FU)/leucovorin/irinotecan/oxaliplatin (mFOLFIRINOX) (6 cycles)
  * Option 2: gemcitabine + nab-paclitaxel (3 cycles)
  * Resectable patients receive surgery 6 weeks post completion of initial chemotherapy
  * Unresectable patients continue with ongoing chemotherapy (option 1 or option 2)
  * Unresectable patients with locoregional progression or metastatic disease, chemotherapy treatment at the discretion of treating medical oncologist
  * Adjuvant chemotherapy for resectable patients to begin within 8 weeks after surgery
  * For patients who received option 1 chemotherapy: 12 weeks of mFOLFIRINOX
  * For patients who received option 2 chemotherapy: 12 weeks of mFOLFIRINOX or 12 additional weeks of gemcitabine/capecitabine
  Interventions: Drug: mFOLFIRINOX; Drug: Gemcitabine + Nab-paclitaxel; Drug: Gemcitabine + Capecitabine; Procedure: Pancreatoduodenectomy (Whipple procedure)
- Arm B (Experimental): * Option 1: fluorouracil(5-FU)/leucovorin/irinotecan/oxaliplatin (mFOLFIRINOX) (6 cycles)
  * Option 2: gemcitabine + nab-paclitaxel (3 cycles)
  * Stereotactic Radiotherapy (SBRT) to commence within 3 weeks of completing initial chemotherapy: 40 Gray (Gy) in 5 fractions over 2 weeks
  * Resectable patients receive surgery 6 weeks post completion of initial chemotherapy
  * Unresectable patients continue with ongoing chemotherapy (option 1 or option 2)
  * Unresectable patients with locoregional progression or metastatic disease, chemotherapy treatment at the discretion of treating medical oncologist
  * Adjuvant chemotherapy for resectable patients to begin within 8 weeks after surgery
  * For patients who received option 1 chemotherapy: 12 weeks of mFOLFIRINOX
  * For patients who received option 2 chemotherapy: 12 weeks of mFOLFIRINOX or 12 additional weeks of gemcitabine/capecitabine
  Interventions: Radiation: Stereotactic Radiotherapy (SBRT); Drug: mFOLFIRINOX; Drug: Gemcitabine + Nab-paclitaxel; Drug: Gemcitabine + Capecitabine; Procedure: Pancreatoduodenectomy (Whipple procedure)

INTERVENTIONS:
Radiation: Stereotactic Radiotherapy (SBRT) — 40 Gray (Gy) in 5 fractions, 2-3 fractions per week over two weeks, 8 Gy per fraction
  Other Names: SBRT; Stereotactic Body Radiotherapy
  Arms: Arm B
Drug: mFOLFIRINOX — * Day 1: oxaliplatin 85mg/m2 + irinotecan 150mg/m2 + leucovorin 50mg
  * 5-FU 2400mg/m2 continuous IV infusion, 46 hour continuous infusion
  * 14-day cycle, 6 cycles
  Other Names: modified regimen of oxaliplatin, leucovorin, irinotecan, and fluorouracil (5-FU)
Drug: Gemcitabine + Nab-paclitaxel — * Day 1, Day 8 and Day 15 gemcitabine 1000mg/m2 + nab-paclitaxel 125mg/m2
  * 28-day cycle, 3 cycles
  Other Names: Gemcitabine + Abraxane
Drug: Gemcitabine + Capecitabine — * Week 1, 2 and 3, qw: 1000 mg/m2 gemcitabine
  * 21 days continuous: 830 mg/m2 oral capecitabine + 7 days rest
  * 28-day cycle, 3 cycles
  Other Names: GemCap
Procedure: Pancreatoduodenectomy (Whipple procedure) — R0 resection. When the tumour is within the head of the pancreas, a standard Whipple's procedure and level 2/3 dissection with modification to obtain margin clearance will be offered. For lesions in the tail, a standard modular resection will be offered.
  Other Names: Whipple

SUMMARY:
This is a prospective, multicentre randomised, phase II clinical trial, with randomisation 2:1 by minimisation and stratification by tumour stage, planned chemotherapy and institution.

DETAILED DESCRIPTION:
This is a prospective, multicentre randomised, phase II clinical trial to evaluate safety and activity of stereotactic body radiotherapy (SBRT) in addition to chemotherapy in patients with high-risk and borderline resectable pancreatic cancer (BRPC) and locally advanced pancreatic cancer (LAPC). High risk defined as any patient with tumour >4cm, extrapancreatic extension or node positive disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged between 18-75 years, with histological confirmation of pancreatic adenocarcinoma
* Any of the following

  1. T3 (tumour >4 cm)
  2. Extrapancreatic extension
  3. Node positive (stage IIB)
  4. Borderline resectable pancreatic cancer, locally advanced pancreatic cancer
* Measurable disease according to RECIST v1.1
* ECOG performance status 0-1
* Adequate renal and haematological function
* Adequate hepatic function. Defined as bilirubin <1.5 X ULN (Upper Limit of Normal), AST + ALT <3.0 X ULN. In patients who have had a recent biliary drainage and whose bilirubin is descending, a value of ≤ 3 X N is acceptable
* Study treatment planned to start within 14 days of registration
* Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments
* Signed, written informed consent

Exclusion Criteria:

* Tumour size greater than 70mm
* Prior abdominal radiotherapy
* Evidence of metastatic disease on baseline radiologic investigations
* History of another malignancy within 2 years prior to randomisation, except adequately treated carcinoma-in-situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial transitional cell carcinoma of the bladder, or any Stage 1 endometrial carcinoma. Patients with a history of other malignancies are eligible if they have been continuously disease free for at least 2 years after definitive primary treatment
* Concurrent illness, including severe infection that may jeopardise the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety
* Neuroendocrine pancreatic carcinoma
* Life expectancy of less than 3 months
* Pregnancy, lactation, or inadequate contraception. Women must be post-menopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration. Men must use a reliable means of contraception
* Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Locoregional control (Locoregional Response Rate LRR) | Within 12 months of randomisation;
  To determine if the addition of SBRT to chemotherapy improves locoregional control;

SECONDARY OUTCOMES:
Safety (NCI CTCAE v5.0) | Safety Assessment before each cycle of chemotherapy, post chemotherapy treatment, following SBRT and surgery (if applicable) then at 3, 6, 9 and 12 months post-randomisation and 6 monthly during year 2, 3 and 4
  Compare acute and late side effects from chemotherapy +/- SBRT
Surgical morbidity/mortality (Clavien grading system) | At discharge post-surgery, 30 days and 90 days post surgery, up to 4 years
  Length of stay, death within 30 days, frequency and severity of adverse events. Hospital admission during surgery will be calculated from day of surgery to date of discharge from acute care hospitalisation. The length of stay in acute hospital care will include intensive care admissions.
Radiological response rates (RECIST v1.1) | at baseline. In SBRT arm, post-initial chemotherapy (prior to SBRT). In both arms, 4-6 weeks post completion of initial treatment (prior to surgery), 3 ,6, 9 and 12 monthly during year 2, 3 and 4.
  Compare radiologic response rates for chemotherapy +/- SBRT
Progression Free Survival (PFS) (RECIST v1.1) | From randomisation to the time of first documented clinical or imaging relapse or date of death from any cause, whichever occurs first; up to 4 years
  Compare 12-month progression free survival
Pathological response rates (College of American Pathology Tumour Regression Grade TRG) | At SRBT/surgery compared to baseline;
  Compare pathologic response rates of chemotherapy +/- SBRT
Surgical resection rates (Guidelines for the Evaluation of Resectability and Histology) | At surgery
  Compare rates of surgical resection
R0 resection rates (>1mm) (Synoptic PC histology reporting as outlined in Royal College of Pathologists of Australasia (RCPA) | At surgery
  Compare R0 resection rates (>1 mm)
Quality of Life (EORTC QLQ C30 and PAN26 QOL) | Baseline, Day 1 of each cycle of chemotherapy, prior to SBRT, post initial chemotherapy +/- SBRT, prior to surgery, 30 days post end of treatment, at months 3, 6,9 and 12 post randomisation 6 monthly in years 2, 3 and 4.
  To assess the impact of the regimens on quality of life of patients
Deterioration-Free Survival (DFS) (EORTC QLQ C30) | The time until the first of the following events: a 10-point deterioration in health status from baseline, disease progression, death, or treatment discontinuation;up to 4 years
  To assess overall net clinical benefit of treatment
Overall Survival (OS) | From the date of randomisation to date of death from any cause, or the date of last known alive; up to 4 years
  OS is defined as the interval from the date of randomisation to date of death from any cause, or the date of last known alive. Participants will be censored at the date of commencement of the subsequent anti-cancer therapy.

OTHER OUTCOMES:
Exploratory biomarker analysis of blood | baseline, prior to SBRT (Arm B only), insertion of fiducial markers (Arm B, optional), post initial treatment, at surgery (optional, at selected sites), 6 and12 months post randomisation and at progression, up to 5 years
  The list of blood biomarkers and their measurement will be updated when confirmed.
Exploratory biomarker analysis of tissue | Diagnosis (archival tissue), at time of fiducial insertion (Arm B, optional), surgical resection (for resectable patients) and at time of progression (optional), up to 5 years.
  The list of tissue biomarkers and their measurement will be updated when confirmed.
ePRO Acceptability | Baseline, Day 1 of each cycle of chemotherapy, 2 weeks post initial chemotherapy(SBRT arm), 4-6 weeks post initial chemotherapy +/- SBRT, 30 days post end of treatment, at months 3, 6,9 and 12 post randomisation 6 monthly in years 2, 3 and 4.
  Proportion of patients who are willing to use electronic device vs. paper format, Analysis of demographic data and assessing data quality between the group

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Oar, Study Chair — ICON Gold Coast University Hospital, Southport, Queensland, AUS
Locations (11):
- Australia (11):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - ICON Cancer Centre, Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
The study will be conducted in accordance with applicable Privacy Acts and Regulations. All data generated in this study will remain confidential. All information will be stored securely at the NHMRC CTC, University of Sydney and will only be available to people directly involved with the study.
  Personal data identifying trial participants will be held securely at the NHMRC CTC for the purpose of follow up if the patient is unable to/wishes to discontinue clinic based follow-up.